CLINICAL TRIAL: NCT01471704
Title: A Phase 1b, Drug-Drug Interaction Study Investigating the Pharmacokinetic Interaction Between INX-08189 and Verapamil HCL ER in Healthy Volunteers
Brief Title: Study Investigating the Pharmacokinetic Interaction Between INX-08189 and Verapamil HCL ER in Healthy Volunteers
Acronym: INX-189-005
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: AI472-005; INH-189-005 (Other: INH-189-005)
Record Dates: First submitted 2011-11-03; First posted 2011-11-16 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Healthy
Keywords: Pharmacokinetics; PK; INX08189; Verapamil; Inhibitex
MeSH Terms: interventions — BMS-986094; Verapamil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- INX-08189 50 mg (Experimental): Study Day 0: Single 50 mg dose of INX-08189 in the morning
  Interventions: Drug: INX-08189 50 mg
- 240 mg verapamil HCL ER (Active Comparator): Study Days 6 to 11: 240 mg verapamil HCL ER once daily (QD) in the morning
  Interventions: Drug: 240 mg verapamil HCL ER
- INX-08189 50 mg & verapamil HCLER 240 mg (Active Comparator): Study Day 12: Co-administration of single 50 mg dose of INX-08189 and 240 mg verapamil HCL ER in the morning
  Interventions: Drug: 50 mg dose of INX-08189 and 240 mg verapamil HCL ER

INTERVENTIONS:
Drug: INX-08189 50 mg — Study Day 0: Single 50 mg dose of INX-08189 in the morning
  Arms: INX-08189 50 mg
Drug: 240 mg verapamil HCL ER — Study Days 6 to 11: 240 mg verapamil HCL ER once daily (QD) in the morning
  Arms: 240 mg verapamil HCL ER
Drug: 50 mg dose of INX-08189 and 240 mg verapamil HCL ER — Study Day 12: Co-administration of single 50 mg dose of INX-08189 and 240 mg verapamil HCL ER in the morning
  Arms: INX-08189 50 mg & verapamil HCLER 240 mg

SUMMARY:
The purpose of this study is to evaluate the potential for a pharmacokinetic (PK) drug-drug interaction between INX-08189 and extended release verapamil hydrochloride (verapamil HCL ER).

DETAILED DESCRIPTION:
This is a single-center, open-label, single-sequence, crossover, drug-drug interaction study in healthy subjects.

Primary Objectives:

Safety

- To evaluate the safety of a single dose of INX-08189 (50 mg) alone and combined with verapamil HCL ER (240 mg) after subjects receive verapamil HCL ER QD for 6 days

Pharmacokinetic

- To evaluate the effect of multiple doses of verapamil HCL ER (240 mg) on the pharmacokinetic (PK) profile of INX-08189 and the metabolite INX-08032, and the effect of a single dose of INX-08189 on the PK profile of verapamil and the metabolite norverapamil

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following criteria at the screening visit (Visit1) and Visit 2 in order to be eligible for study drug administration:

1. Must be a healthy male or female between 18 and 55 years of age (inclusive) with body mass index (BMI) between 18 and 30 kg/m2 (inclusive), and weigh > 50 kg at the time of signing the informed consent;
2. Capable of giving written informed consent that includes compliance with the requirements and restrictions listed in the consent form. Signed informed consent must be on file prior to screening procedures;
3. Subject is able to understand and comply with the protocol requirements, instructions and restrictions;
4. Must be a non-tobacco user for at least 3 months prior to selection;
5. Healthy on the basis of physical examination, medical history, vital signs, electrocardiogram and clinical laboratory tests at screening;
6. Women must be postmenopausal for at least 2 years or be surgically sterile with complete hysterectomy or bilateral oophorectomy, and not be pregnant nor be breastfeeding;
7. Male subjects, who are not surgically sterile with vasectomy, must agree to use a double barrier method of birth control, such as, a condom plus spermicidal agent (foam/gel/film/cream/suppository). This criterion must be followed from the time of the first dose of study medication until 30 days after the last dose of medication. Male subjects cannot donate sperm during the study and for 3 months after receiving the last dose of the study drug.

Exclusion Criteria:

Subjects must NOT meet the following criteria at the Screening Visit (Visit1), in order to be eligible for study drug administration at Visit 2:

1. Infection with Hepatitis A, B or C Virus;
2. Infection with the Human Immunodeficiency Virus (HIV);
3. History of or any current medical condition which could impact the safety of the participant in the study;
4. Current active or underlying GI, cardiovascular, neurologic, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory, or infectious disease;
5. Clinically significant abnormalities on centrally read ECG including evidence of bradycardia (rate < 60 bpm) or evidence of PR prolongation;
6. Screening vital signs representing a heart rate of < 60 bpm, systolic blood pressure < 90 mm Hg, and diastolic blood pressure < 60 mm Hg;
7. Currently significant diarrhea, gastric stasis, or constipation that in the investigator's opinion could influence drug absorption or bioavailability;
8. Safety laboratory abnormalities at screening which are clinically significant, or absolute neutrophil count of < 1800 cells/mm3, or platelet count < 130,000 cells/mm3, or hemoglobin < 12 g/dl for women and < 13 g/dl for men;
9. Women of child bearing potential, pregnant or breastfeeding;
10. Current abuse of alcohol or illicit drugs, or history of alcohol or illicit drug abuse within the preceding 2 years;
11. A positive urine drug test at screening;
12. Consumption of more than 2 units of alcoholic beverages per day or more than 14 units per week (1 unit of alcohol equals 1 glass of beer, 1 glass of wine, 25ml shot of 40% spirit), consumption of alcohol 72 hours before or after study medication intake, consumption of an average of more than five (5) 240 ml servings of coffee or other caffeinated beverages per day;
13. Use of chronic prescription medications within 3 months, acute prescription medications within 14 days, or systemic over-the-counter (OTC) medications, including vitamins, within 7 days of starting the study;
14. Received an investigational drug or vaccine or used an investigational medical device within 3 months or 5 half lives (whichever is longer) before the planned start of treatment or having participated previously in a study with INX-08189;
15. Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 28 days prior to the first dose and throughout the study;
16. Consumption of grapefruit or grapefruit juice starting 48 hours before Study Day -1, during the subject's confinement in the unit, and during the outpatient follow-up periods.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Effect of multiple doses of verapamil HCL ER 240 mg on the PK profile of INX-08189, and the effect of a single dose of INX-08189 on the PK profile of verapamil. | INX-08189 and Verapamil: Study Day 0 (INX-08189), Study Day 12 (Verapamil) and subsequently at 30 minutes, and 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 hours after dosing. INX-08189 also at 48, 72, and 96 hours after initial dose.
  PK for INX-08189 and verapamil by: maximum plasma concentration (Cmax), time Cmax is observed (Tmax), plasma concentration at end of dosing (Ctau), area under plasma concentration-time curve; time 0 to last measurable plasma concentration (AUC0-last), area under plasma concentration-time curve; time 0 to infinity (AUC0-inf), area under plasma concentration-time curve; 0 to end of dosing (AUC0-tau), elimination half-life (t1/2), apparent oral clearance (CL/F), and apparent oral volume of distribution (Vz/F).
Safety of a single dose of INX-08189 50 mg alone & combined with verapamil HCL ER 240 mg after subjects received verapamil HCL ER QD for 6 days | Study Day -1, during the 24-hours post-dose, Study Day 2 to 4, 5, 6, 7 to 11, 12, and 13 to 16
  Safety and tolerability parameters, including adverse event, concurrent medication, clinical laboratory, electrocardiogram (ECG) and vital signs assessments

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Campaneria, MD, Study Director
Locations (1):
- Prism Research, LLC, Saint Paul, Minnesota, United States